CLINICAL TRIAL: NCT01554163
Title: A Phase III, 12-Week, Randomized, Active-Comparator-Controlled, Parallel-Group, Double Blind Study in Korea to Assess the Safety and Efficacy of Etoricoxib 30 mg Versus Celecoxib 200 mg in Patients With Osteoarthritis
Brief Title: Safety and Efficacy of Etoricoxib 30 mg Versus Celecoxib 200 mg in Korean Participants With Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0663-112
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Celecoxib; Etoricoxib
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Etoricoxib; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etoricoxib 30 mg (Experimental): Etoricoxib, 30 mg tablet, orally, once daily for 12 weeks.
  Interventions: Drug: Etoricoxib 30 mg
- Celecoxib 200 mg (Active Comparator): Celecoxib, 200 mg capsule, orally, once daily for 12 weeks.
  Interventions: Drug: Celecoxib 200 mg

INTERVENTIONS:
Drug: Etoricoxib 30 mg — Etoricoxib 30 mg tablet once daily for 12 weeks.
  Other Names: MK-0663; Arcoxia
  Arms: Etoricoxib 30 mg
Drug: Celecoxib 200 mg — Celecoxib 200 mg once daily for 12 weeks
  Other Names: Celebrex; Celebra
  Arms: Celecoxib 200 mg

SUMMARY:
The main purpose of this study is to establish that etoricoxib 30 mg is safe and not inferior to celecoxib 200 mg in the treatment of the signs and symptoms of osteoarthritis in Korean patients. Given that the efficacy of etoricoxib vs. placebo in the treatment of osteoarthritis has been established, and that prescription drugs, such as celecoxib, are available for the treatment of pain associated with osteoarthritis in Korea, it would be inappropriate to subject patients with a flare of osteoarthritic pain to the placebo treatment for 12 weeks, and thus the study is designed as an active-comparator study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 40 years of age
* Clinical diagnosis of osteoarthritis of the knee for greater than 6 months based on clinical and radiographic criteria
* Female patients of childbearing potential must have a negative pregnancy test prior to study enrollment and must agree to remain abstinent, and use barrier, intramuscular, or implanted contraceptives from Visit 1 until 28 days after the last dose of study medication.
* Patient is of American Rheumatism Association (ARA) functional Class I, II, or III
* Patient is willing to limit alcohol intake to 2 or less drinks per day during study and the follow-up period
* Patient is willing to avoid unaccustomed physical activity for the duration of the study and follow-up period
* With the exception of osteoarthritis, the patient is judged to be in good general health based on medical history, physical exam, and routine laboratory tests
* Patient is able to read, understand and complete study questionnaires, including questions requiring a visual analog scale (VAS) response
* Patient provides written informed consent for the trial
* For prior non-steroidal anti-inflammatory drug (NSAID) users only, the patient has a history of positive therapeutic benefit with NSAIDs and has taken an NSAID prior to study enrollment and at a therapeutic dose level prior to study enrollment (Visit 1)
* For prior NSAID users only, the patient assessment of Pain Walking on a Flat Surface (WOMAC Section A, Question1) at Visit 1 (prestudy) is less than 80 mm (100 mm VAS)
* For prior NSAID users only, prior to randomization, and following discontinuation of NSAIDs during the washout period specified patients must satisfy the following 3 flare criteria: Minimum of 40 mm on patient reported Pain Walking on a Flat Surface (WOMAC Section A, Question 1); Increase of 15 mm on patient reported Pain Walking on a Flat Surface (WOMAC Section A, Question 1) compared to prestudy baseline recorded at Visit 1; and A worsening in Investigator Global Assessment of Disease Status of at least 1 category on a 5 category scale compared to Visit 1 recording
* For prior acetaminophen/paracetamol users only, patient has taken acetaminophen/paracetamol on a regular basis prior to study enrollment (Visit 1) and does not use NSAIDs for the treatment of osteoarthritis of the knee
* For prior acetominophen/paracetamol users only, at both Visits 1 and 2, patients must satisfy all of the following 3 criteria: Minimum of 40 mm on patient reported Pain Walking on a Flat Surface (WOMAC Section A, Question 1); Investigator Global Assessment of Disease Status as fair, poor, or very poor; and Minimum of 40 mm on Patient Global Assessment of Disease Status (100 mm

VAS)

Exclusion Criteria:

* Patient has a concurrent medical/arthritic disease that could confound or interfere with evaluation of efficacy
* Patient is legally incompetent (e.g., a minor or mentally incapacitated), or has active psychosis, or significant emotional problems at the time of the study which in the view of the investigator are sufficient to interfere with the conduct of the study
* Patient has a history of gastric or biliary surgery (including gastric bypass surgery), or small intestine surgery that causes clinical malabsorption
* Patient is allergic to, or has a history of a significant clinical or laboratory adverse experience associated with etoricoxib or celecoxib or any of their constituents
* Patient is allergic to acetaminophen/paracetamol, or has hypersensitivity (e.g., bronchoconstriction in association with nasal polyps) to aspirin or NSAIDs
* Patient has an estimated glomerular filtration rate is less than or equal to 30 ml/min
* Patient has Class II-IV congestive heart failure
* Patient has established ischemic heart disease, cerebrovascular disease, or peripheral vascular disease
* Patient has uncontrolled hypertension with an diastolic exclusionary limit of > 90 mm Hg and a systolic exclusionary limit of > 140 mm Hg
* Patient has moderate or severe hepatic insufficiency defined as Child Pugh score > 6
* Patient has a history of neoplastic disease
* Patient has a history of any illness, which in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient
* Patient is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within the last 5 years) of drug or alcohol abuse or dependence
* Patients considered morbidly obese with a body mass index (BMI) ≥ 35 kg/m^2
* Patient has new use (within 2 weeks of Visit 1 and during the entire duration of the study and follow-up period) of physical medicine modalities involving the study joint, including but not limited to: physical therapy, chiropractic interventions, acupuncture, Transcutaneous Electrical Nerve Stimulator (TENS), and ultrasound
* Patient is expected to undergo surgery involving the study joint during the course of the study
* Patients taking oral contraceptives
* Patients using intra-articular steroids or hyaluronic acid injections to the study knee or other immunosuppressant medication within 3 months of Visit 1
* Patients using intravenous, intramuscular, or oral corticosteroids, intra-articular steroids or hyaluronic acid injections to any joint other than the study joint within 1 month of Visit 1
* Patients using topical or systemic analgesic medications within 3 days of Visit 1 and throughout the duration of the study
* Patients using non-study NSAID or cyclooxygenase 2 (COX-2) specific inhibitor during the study treatment period, with the exception of low-dose aspirin (≤ 325 mg/day)
* Patients receiving a Chinese traditional arthritis treatment within 1 week of Visit 1
* Patients with clinically significant abnormalities on Visit 1 clinical examination or laboratory safety tests. Serum transaminases should be ≤ 150% of the upper limit of normal
* Patients currently participating in or has participated in a study with an

investigational drug or device within 4 weeks of signing informed consent

* Patients with an active peptic ulcer or a history of inflammatory bowel disease
* Patients with a personal or family history of an inherited or acquired bleeding
* Patients that are pregnant or breast-feeding, or expecting to conceive within the projected duration of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

REFERENCES:
- [Result] Yoo MC, Yoo WH, Kang SB, Park YW, Kim SS, Moon KH, Song YW, Min BW, Cho YJ, Moon SH, Bin SI, Baek HJ, Shim SC, Lee SW, Yoo DH, Mehta A, Skuban A, Cukrow DM, Vandormael K, Yan L. Etoricoxib in the treatment of Korean patients with osteoarthritis in a double-blind, randomized controlled trial. Curr Med Res Opin. 2014 Dec;30(12):2399-408. doi: 10.1185/03007995.2014.955169. Epub 2014 Sep 3. PMID 25133963

RESULTS

PARTICIPANT FLOW:
Groups:
- Etoricoxib 30 mg: Etoricoxib 30 mg administered orally once daily for 12 weeks.
- Celecoxib 200 mg: Celecoxib 200 mg administered orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Etoricoxib 30 mg | Celecoxib 200 mg
Started | 120 | 119
Number Treated | 119 | 119
Completed | 112 | 109
Not Completed | 8 | 10
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-Compliance With Study Drug | 1 | 1
Not completed — Protocol Violation | 0 | 4
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etoricoxib 30 mg | Celecoxib 200 mg | Total
Number analyzed (Participants) | 120 | 119 | 239
Age, Customized [Number; unit: Participants]
  40 to 50 years | 4 | 10 | 14
  51 to 60 years | 41 | 40 | 81
  61 to 70 years | 46 | 47 | 93
  71 to 80 years | 27 | 18 | 45
  81 to 90 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 104 | 214
  Male | 10 | 15 | 25

OUTCOME MEASURES:

1. Primary Outcome: Time-Weighted Mean Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale
Description: The WOMAC osteoarthritis scale consists of 24 items in 3 subscales: pain, stiffness, and physical function. The pain subscale rates participant pain during walking, using stairs, in bed, sitting or lying, and standing using a visual analog scale (VAS) from 0-100mm where 0 is the best possible level of pain and 100 is the highest level of pain. The pain subscale is calculated as the average of the responses to the 5 questions related to pain. The calculation of the time-weighted average was done by taking the time between adjacent observations divided by the time from the randomization visit to the last observation in the period of interest, and using it as the weight for computation of the average.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: The population consisted of all participants that received one dose of study medication and had a baseline value for the WOMAC pain subscale, and had at least one post-randomization observation.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 30 mg | Celecoxib 200 mg
Number analyzed (Participants) | 119 | 119
Score on a Scale | -21.40 (1.35) | -19.76 (1.34)
Statistical Analysis 1: Comparison: Etoricoxib 30 mg vs Celecoxib 200 mg; Test type: Non-Inferiority or Equivalence — Etoricoxib 30 mg will be considered non-inferior to celecoxib 200 mg if the upper bound of the two-sided 95% confidence interval of the betweentreatment difference in LS mean time-weighted average change from baseline over 12 weeks in WOMAC Pain Subscale (VAS) is no greater than 10 mm (non-inferiority margin); p = 0.390, ANCOVA; Difference in LS Mean Change = -1.63, 95% CI 2-sided [-5.37 to 2.10]

2. Secondary Outcome: Time-Weighted Mean Change From Baseline in the WOMAC Physical Function Subscale
Description: The WOMAC osteoarthritis scale consists of 24 items in 3 subscales: pain, stiffness, and physical function. The physical function subscale rates participant pain during stair use, rising from sitting, standing, bending, walking, getting in/out of a car, shopping, putting on/taking off socks, rising from bed, lying in bed, getting in/out of the bath, sitting, getting on/off the toilet, heavy household duties, and light household duties using a visual analog scale (VAS) from 0-100mm where 0 is the best possible level of functioning and 100 is the highest level of functioning. The physical function subscale was calculated as the average of the responses to the 17 questions related to functional status. The calculation of the time-weighted average was done by taking the time between adjacent observations divided by the time from the randomization visit to the last observation in the period of interest, and using it as the weight for computation of the average.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: The population consisted of all participants that received one dose of study medication and had a baseline value for the WOMAC physical function subscale, and had at least one post-randomization observation.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 30 mg | Celecoxib 200 mg
Number analyzed (Participants) | 119 | 119
Score on a Scale | -17.78 (1.28) | -16.46 (1.28)
Statistical Analysis 1: Comparison: Etoricoxib 30 mg vs Celecoxib 200 mg; Test type: Non-Inferiority or Equivalence — Etoricoxib 30 mg will be considered non-inferior to celecoxib 200 mg if the upper bound of the two-sided 95% confidence interval of the between-treatment difference in LS means (etoricoxib minus celecoxib) is no greater than 10 mm; p = 0.464, ANCOVA; Difference in LS Mean Change = -1.32, 95% CI 2-sided [-4.88 to 2.23]

3. Secondary Outcome: Time-Weighted Mean Change From Baseline in the Participant Global Assessment of Disease Status
Description: The Participant Global Assessmet of Disease was a one item questionnaire that asked participants to answer the following question, "Considering all the ways your arthritis affects you, mark (X) on the scale for how well you are doing." The questionnaire employed a 0-100 mm visual analog scale (VAS) to record participant responses, with 0 representing the best possible assessment and 100 representing the worst possible assessment. The calculation of the time-weighted average was done by taking the time between adjacent observations divided by the time from the randomization visit to the last observation in the period of interest, and using it as the weight for computation of the average.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: The population consisted of all participants that received one dose of study medication and had a baseline value for the Participant Global Assessment of Disease Status, and had at least one post-randomization observation.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 30 mg | Celecoxib 200 mg
Number analyzed (Participants) | 119 | 119
Score on a Scale | -24.71 (1.58) | -23.61 (1.58)
Statistical Analysis 1: Comparison: Etoricoxib 30 mg vs Celecoxib 200 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.624, ANCOVA; Difference in LS Mean Change = -1.09, 95% CI 2-sided [-5.48 to 3.30]

4. Secondary Outcome: Time-Weighted Mean Response in the Participant Global Assessment of Response to Therapy
Description: Participants were asked to rate their global assessment of response to therapy on a Likert scale from 0 to 4, with 0 = excellent, 1 = good, 2 = fair, 3 = poor, 4 = none. The calculation of the time-weighted average was done by taking the time between adjacent observations divided by the time from the randomization visit to the last observation in the period of interest, and using it as the weight for computation of the average.
Time Frame: Week 2, Week 6, Week 12
Population: The population consisted of all participants that received one dose of study medication and had a Week 2, Week 6, and Week 12 value for the Participant Global Assessment of Response to Therapy.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 30 mg | Celecoxib 200 mg
Number analyzed (Participants) | 119 | 119
Score on a Scale | 1.48 (0.06) | 1.56 (0.07)
Statistical Analysis 1: Comparison: Etoricoxib 30 mg vs Celecoxib 200 mg; Test type: Superiority or Other; p = 0.369, ANCOVA; Difference in LS Mean Change = -0.08, 95% CI 2-sided [-0.26 to 0.10]

5. Secondary Outcome: Time-Weighted Mean Change From Baseline in the Investigator Global Assessment of Disease Status
Description: Study investigators were asked to rate the global assessment of participant disease status on a Likert scale from 0 to 4, with 0 = very well, 1 = good, 2 = fair, 3 = poor and 4 = very poor. The calculation of the time-weighted average was done by taking the time between adjacent observations divided by the time from the randomization visit to the last observation in the period of interest, and using it as the weight for computation of the average.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: The population consisted of all participants that received one dose of study medication and had a baseline value for the Investigator Global Assessment of Disease Status, and had at least one post-randomization observation.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 30 mg | Celecoxib 200 mg
Number analyzed (Participants) | 119 | 119
Score on a Scale | -1.71 (0.06) | -1.62 (0.06)
Statistical Analysis 1: Comparison: Etoricoxib 30 mg vs Celecoxib 200 mg; Test type: Superiority or Other; p = 0.294, ANCOVA; Difference in LS Mean Change = -0.09, 95% CI 2-sided [-0.25 to 0.08]

6. Secondary Outcome: Time-Weighted Mean Change From Baseline in the WOMAC Stiffness Subscale
Description: The WOMAC osteoarthritis scale consists of 24 items in 3 subscales: pain, stiffness, and physical function. The stiffness subscale rates stiffness after first waking and later in the day using a visual analog scale (VAS) from 0-100mm where 0 is the best possible level of stiffness and 100 is the highest level of stiffness. The stiffness subscale is calculated as the average of the responses to the 2 questions related to stiffness. The calculation of the time-weighted average was done by taking the time between adjacent observations divided by the time from the randomization visit to the last observation in the period of interest, and using it as the weight for computation of the average.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: The population consisted of all paricipants that received one dose of study medication and had a baseline value for the WOMAC stiffness subscale, and had at least one post-randomization observation.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 30 mg | Celecoxib 200 mg
Number analyzed (Participants) | 119 | 119
Score on a Scale | -18.41 (1.48) | -17.55 (1.48)
Statistical Analysis 1: Comparison: Etoricoxib 30 mg vs Celecoxib 200 mg; Test type: Superiority or Other; p = 0.679, ANCOVA; Difference in LS Mean Change = -0.86, 95% CI 2-sided [-4.96 to 3.24]

7. Secondary Outcome: Time-Weighted Mean Response on the Investigator Global Assessment of Response to Therapy
Description: Study investigators were asked to rate the global assessment of participant response to therapy on a Likert scale from 0 to 4, with 0 = excellent, 1 = good, 2 = fair, 3 = poor, 4 = none. The calculation of the time-weighted average was done by taking the time between adjacent observations divided by the time from the randomization visit to the last observation in the period of interest, and using it as the weight for computation of the average.
Time Frame: Week 6, Week 12
Population: The population consisted of all participants that received one dose of study medication and had a value at Week 6 and Week 12 for the Investigator Global Assessment of Response to Therapy.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Etoricoxib 30 mg | Celecoxib 200 mg
Number analyzed (Participants) | 119 | 119
Score on a Scale | 1.39 (0.07) | 1.49 (0.07)
Statistical Analysis 1: Comparison: Etoricoxib 30 mg vs Celecoxib 200 mg; Test type: Superiority or Other; p = 0.314, ANCOVA; Difference in LS Mean Change = -0.10, 95% CI 2-sided [-0.30 to 0.10]

ADVERSE EVENTS:
Time Frame: Up to 12 weeks.
Arm/Group | Etoricoxib 30 mg | Celecoxib 200 mg
Serious Adverse Events (participants affected / at risk) | 0/119 | 1/119
Other Adverse Events (participants affected / at risk) | 12/119 | 3/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib 30 mg (N=119) | Celecoxib 200 mg (N=119)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib 30 mg (N=119) | Celecoxib 200 mg (N=119)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (20) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.